CLINICAL TRIAL: NCT06646952
Title: CD147 Targeting Nanobody Probe for PET Imaging in Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Hua Zhu (Other)
Responsible Party: Sponsor-Investigator, Hua Zhu, Principal Investigator, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Other Study IDs: 2024KT10
Record Dates: First submitted 2024-10-10; First posted 2024-10-17 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor
Keywords: CD147; solid tumor
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-NOTA-MAL-NB147: All enrolled participants will be allocated to this arm (single-arm study). Study participants will undergo 68Ga-NOTA-MAL-NB147 PET/CT scan.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/ CT scan.

SUMMARY:
The objective of the study is to construct a noninvasive approach using 68Ga-NOTA-MAL-NB147 PET/CT to detect the CD147 expression of tumor lesions in patients with Solid tumors and to identify patients benefiting from CD147 targeting treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or cytologically confirmed malignant melanoma, hepatocellular carcinoma, colorectal cancer, pancreatic cancer, breast cancer, gastric cancer, and lung cancer.
2. Aged ≥18 and ≤75 years, with no gender restrictions.
3. ECOG score of 0 or 1.
4. Expected survival time ≥6 months.
5. At least one easily accessible lesion that can be biopsied within one month before or after the PET scan. The patient consents to using archived or fresh biopsy tissue samples for relevant analysis.
6. Blood routine and liver/kidney function must meet the following criteria: Blood routine: WBC ≥ 4.0×10⁹/L or neutrophils ≥ 1.5×10⁹/L, PLT ≥ 100×10⁹/L, Hb ≥ 90 g/L; PT or APTT ≤ 1.5 ULN; Liver/kidney function: T-Bil ≤ 1.5×ULN (upper limit of normal), ALT/AST ≤ 2.5×ULN or 5×ULN (for subjects with liver metastases), ALP ≤ 2.5×ULN (if bone or liver metastases exist, ALP ≤ 4.5×ULN); BUN ≤ 1.5×ULN; SCr ≤ 1.5×ULN; At least one measurable target lesion according to RECIST 1.1 criteria.
7. Women must use contraceptive measures during the study or for six months after the study ends (effective contraceptive methods include sterilization, hormonal intrauterine devices, condoms, contraceptive pills/devices, abstinence, or partner tubal ligation, etc.). Men must agree to use contraceptive measures during the study or for six months after the study ends.
8. Able to understand and voluntarily sign the informed consent form, with good compliance.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning to become pregnant during the study or within three months after administration, as well as individuals donating sperm or oocytes.
2. Individuals known or suspected to be allergic to the investigational drug or any of its components.
3. Individuals with significantly abnormal liver or kidney function: serum total bilirubin (TBIL) > 1.5 × 20 µmol/L, or aspartate aminotransferase (AST) > 2.5 × 45 µmol/L, or alanine aminotransferase (ALT) > 2.5 × 40 µmol/L, or serum creatinine > 1.5 × 130 µmol/L.
4. Unable to cooperate in completing the PET scan, or suffering from claustrophobia or other conditions that prevent cooperation during the PET scan.
5. Other situations deemed inappropriate for participation in the trial by the investigator. Female patients who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Malignant tumor patients or suspected patients
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions。 The uptake of the tracer （68Ga-NOTA-MAL-NB147） in solid tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No